CLINICAL TRIAL: NCT02984631
Title: The Evaluation and Treatment of Elevated Left-Sided Filling Pressures by Balloon Inflation Within the Interior Vena Cava
Brief Title: The Evaluation and Treatment of Elevated Left-Sided Filling Pressures by Balloon Inflation Within the IVC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cardioflow Technologies, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CFT-37215-ECH-02
Record Dates: First submitted 2016-12-03; First posted 2016-12-07 (Estimated); Last update posted 2018-04-09 (Actual); Status verified 2018-04

CONDITIONS: Hypertension, Pulmonary; Heart Failure
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preventing pulm HTN during exercise 2nd (Other): Standard of care invasive cardiopulmonary exercise test (CPET) followed by CPET with pre-load control.
  Interventions: Procedure: Preventing pulm HTN during exercise
- Preventing pulm HTN during exercise 1st (Other): Pre-load control of invasive cardiopulmonary exercise test (CPET) followed by standard CPET.
  Interventions: Procedure: Preventing pulm HTN during exercise

INTERVENTIONS:
Procedure: Preventing pulm HTN during exercise — Balloon catheter is inflated within the IVC to maintain pulmonary pressures during exercise.

SUMMARY:
In patients with heart failure, elevated filling pressures may contribute to symptoms while not improving cardiac output. The current study is focused on evaluating the relationship between exercise capacity, pulmonary pressures, cardiopulmonary parameters, and symptoms of dyspnea in patients with heart failure during exercise.

DETAILED DESCRIPTION:
Previous studies have suggested that intracardiac pressures can be decreased without compromising cardiac function. During an invasive cardiopulmonary exercise test (CPET), catheters are placed within the heart and pulmonary vasculature to evaluate cardiopulmonary function in response to exercise. We will be testing whether pulmonary hypertension can be prevented during exercise by adjusting right ventricular pre-load. We will also be evaluating parameters of cardiopulmonary function during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects scheduled to undergo an exercise right heart catheterization at El Camino Hospital.
2. New York Heart Association (NYHA) II or III.
3. Subjects must be between 18 and 80 years of age.
4. A left ventricular ejection fraction ≥ 35%.
5. Subjective or objective evidence (e.g. 6 minute walk test) of impaired exercise capacity.
6. Is willing and able to sign an IRB-approved written informed consent

Exclusion Criteria:

1. Inability to peddle exercise while laying flat.
2. More than mild valve disease.
3. Clinical or objective evidence of inducible myocardial ischemia.
4. Significant lung disease, such as prior diagnosis of COPD.
5. Resting or dynamic outflow tract gradient.
6. Severe pulmonary HTN (>60mmHg at rest)
7. Moderate to severe RV dysfunction
8. History of DVT, PE
9. Pregnancy (women of child-bearing age, regardless of contraceptive measures, must be willing to take a pregnancy test prior to the study).
10. Recent major surgery or hospitalization (within 30 days)
11. Participation in another clinical study (within 30 days)
12. Advanced neurological disease (e.g. dementia)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12 (Actual); Primary Completion 2019-06 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Reduction in respiratory rate at matched levels of exercise. | During the CPET, within 30 minutes of study.

SECONDARY OUTCOMES:
Change in patient symptoms-- dyspnea and leg discomfort (Borg units) | During the CPET, within 30 minutes of study.
Change in ventilatory threshold | During the CPET, within 30 minutes of study.
Change in exercise time | During the CPET, within 30 minutes of study.
Change in heart rate for given level of exercise (work rate in watts) | During the CPET, within 30 minutes of study.
Change in anaerobic threshold | During the CPET, within 30 minutes of study.
Change in pulmonary diastolic pressure for a given level of exercise (work rate) | During the CPET, within 30 minutes of study.
Change in dead space ventilation at a given level of exercise (and VE/VCO2 slope) | During the CPET, within 30 minutes of study.
Change in cardiac output at a given level of exercise | During the CPET, within 30 minutes of study.
Determining predictors of peak VO2 | During the CPET, within 30 minutes of study.
Change in oxygen uptake at a given level of exercise | During the CPET, within 30 minutes of study.
Change in pH level at a given level of exercise | During the CPET, within 30 minutes of study.
Change in Peak VO2 | During the CPET, within 30 minutes of study.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Kaiser, MD, Principal Investigator — Electrophysiologist at El Camino Hospital.
Locations (1):
- El Camino Hospital, Mountain View, California, United States

IPD SHARING:
Plan to Share IPD: Undecided